CLINICAL TRIAL: NCT01431521
Title: An Exploratory Study to Evaluate Changes in Hepatic Fat Following Multiple-Dose Administration of MK-4074 and Pioglitazone Hydrochloride
Brief Title: Study of Changes in Hepatic Fat Following Administration of MK-4074 and Pioglitazone Hydrochloride (MK-4074-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4074-008
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-4074 (Experimental): Participants will receive oral doses of MK-4074 200 mg (2 x 100-mg capsules) twice daily for 4 weeks.
  Interventions: Drug: MK-4074 200 mg
- Placebo for MK-4074 (Placebo Comparator): Participants will receive oral doses of placebo to match MK-4074 twice daily for 4 weeks.
  Interventions: Drug: Placebo for MK-4074
- Pioglitazone (Experimental): Participants will receive oral doses of pioglitazone hydrochloride 30 mg (1 x 30-mg tablet) once daily for 4 weeks.
  Interventions: Drug: Pioglitazone hydrochloride 30 mg
- Placebo for pioglitazone (Placebo Comparator): Participants will receive oral doses of placebo to match pioglitazone hydrochloride once daily for 4 weeks.
  Interventions: Drug: Placebo for pioglitazone hydrochloride

INTERVENTIONS:
Drug: MK-4074 200 mg — 2 x 100-mg capsules, orally, twice-daily (BID) for 4 weeks
  Arms: MK-4074
Drug: Placebo for MK-4074 — 2 x 100-mg capsules, orally, BID for 4 weeks.
  Arms: Placebo for MK-4074
Drug: Pioglitazone hydrochloride 30 mg — 1 x 30-mg tablet, orally, once daily for 4 weeks
  Arms: Pioglitazone
Drug: Placebo for pioglitazone hydrochloride — 1 x 30-mg tablet, orally, once daily for 4 weeks
  Arms: Placebo for pioglitazone

SUMMARY:
This study will evaluate changes in liver fat content following multiple oral doses of MK-4074 and Pioglitazone Hydrochloride in adult males and females with fatty liver disease. The primary hypothesis of the study is that a multiple-dose administration of MK-4074 200 mg twice daily for 4 weeks results in a decrease in hepatic fat content with respect to placebo in adult male and female participants with hepatic steatosis (i.e., on order of 50% reduction in hepatic fat with respect to placebo is expected).

ELIGIBILITY:
Inclusion Criteria:

* Females must be of non-childbearing potential
* Body mass index (BMI) ≥32.0 kg/m^2
* In good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests
* No clinically significant abnormality on electrocardiogram
* Has documented hepatic fat content ≥10% within 6 months of enrollment
* Maintained stable weight (by history) for at least 4 weeks
* Agrees not to initiate a weight loss program and agrees to maintain consistent dietary habits and exercise routines for the duration of the study
* Has a rating of 'moderate' or 'severe' steatosis on ultrasound at the prestudy (screening) visit

Exclusion Criteria:

* Change in weight greater than 4% between prestudy visit and randomization into the study
* History of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant
* Liver disease other than fatty liver or non-alcoholic steatohepatitis (NASH)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3x the upper limit of normal range
* Serum triglyceride level >600 mg/dL
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular (including congestive heart failure), hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Had abdominal surgery, gastric bypass, bowel resection, recent liver biopsy, or any other procedure within a minimum of 4 weeks
* History of neoplastic disease
* Claustrophobia or other contraindication to magnetic resonance imaging (MRI)
* Have not washed off agents associated with changes in hepatic fat or used for treatment of Non-alcoholic fatty liver disease (NAFLD) or NASH for a minimum of 3 months prior
* Consumes excessive amounts of alcohol, coffee, tea, cola, or other caffeinated beverages
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks
* Significant multiple and/or severe allergies
* Intolerance or hypersensitivity to pioglitazone hydrochloride or any inactive ingredients
* Regular user of any illicit drugs or has a history of drug (including alcohol) abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-26 (Actual); Primary Completion 2012-09-18 (Actual); Study Completion 2012-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4074-008&kw=4074-008&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one male or female participants (non-childbearing potential) between the ages of 18 and 60, inclusive, with body mass index (BMI) ≥ 32 kg/m^2 were enrolled in the study. Participants were pre-screened by means of ultrasound, and only those participants with a rating of "moderate" or "severe" steatosis were further evaluated by means of MRI.
Period: Overall Study
Arm/Group | MK-4074 | Placebo for MK-4074 | Pioglitazone | Placebo for Pioglitazone
Started | 10 | 5 | 11 | 5
Treated | 10 | 5 | 10 | 5
Completed | 10 | 5 | 10 | 5
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-4074 | Placebo for MK-4074 | Pioglitazone | Placebo for Pioglitazone | Total
Number analyzed (Participants) | 10 | 5 | 11 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (5.8) | 48.0 (7.6) | 43.7 (12.1) | 47.8 (10.6) | 42.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 4 | 7
  Male | 10 | 4 | 9 | 1 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Hepatic Fat
Description: Hepatic fat content was assessed via magnetic resonance imaging (MRI) prior to first dose administration and following 4 weeks of treatment. Percent change in hepatic fat fraction from baseline was calculated for each of the 9 liver regions separately and then these were averaged to calculate overall percent change from baseline for each participant.
Time Frame: Baseline and Week 4
Population: Per-Protocol (PP) Population consists of those participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo: Participants will receive oral doses of placebo to match MK-4074 or pioglitazone hydrochloride once daily for 4 weeks.
Arm/Group | MK-4074 | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Percent change | -35.73 [-44.53 to -26.93] | -18.04 [-26.84 to -9.24] | 8.63 [-0.17 to 17.43]
Statistical Analysis 1: Comparison: MK-4074 vs Placebo; Test type: Superiority or Other; p < 0.001, Linear mixed effects model; Treatment as fixed factor and predose Day 1 value, as a fixed covariate; Least squares mean difference = -44.37, 95% CI 2-sided [-54.67 to -34.07]
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p < 0.001, Linear mixed effects model; Treatment as fixed factor and predose Day 1 value, as a fixed covariate; Least squares mean difference = -26.67, 95% CI 2-sided [-36.97 to -16.37]
Statistical Analysis 3: Comparison: MK-4074 vs Pioglitazone; Test type: Superiority or Other; p = 0.007, Linear mixed effects model; Treatment as fixed factor and predose Day 1 value, as a fixed covariate; least squares mean difference = -17.69, 95% CI 2-sided [-36.97 to -7.39]

2. Secondary Outcome: Percent Change From Baseline in Alanine Transaminase (ALT)
Description: Hepatic steatosis is not uncommonly associated with mild elevations in serum transaminases, specifically ALT, and these elevations may be a marker of more advanced hepatic disease. Serum transaminases were monitored at baseline and once weekly for the duration of the study to permit a better understanding of the time course of potential improvement in hepatic inflammation during the course of this short study.
Time Frame: Baseline and Week 4
Population: The AST Population consists of all participants who received at least one dose of the study drug. One participant in the Placebo group did not have ALT data for Day 28.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | MK-4074 | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 10 | 9
Percent change | -9.82 [-21.13 to 1.49] | -20.21 [-31.52 to -8.90] | -3.47 [-15.08 to 8.13]
Statistical Analysis 1: Comparison: MK-4074 vs Placebo; Test type: Superiority or Other; p > 0.200, Linear mixed effect model; Containing fixed effects for treatment, and predose Day 1 (baseline) as a fixed covariate; Least square mean difference = -6.35, 95% CI 2-sided [-18.69 to 6.00]
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.028, Linear mixed effects model; Containing fixed effects for treatment, and predose Day 1 (baseline) as a fixed covariate; Least squares mean difference = -16.74, 95% CI 2-sided [-29.08 to -4.40]

3. Secondary Outcome: Percent Change From Baseline Aspartate Transaminase (AST)
Description: Hepatic steatosis is not uncommonly associated with mild elevations in serum transaminases, including AST, and these elevations may be a marker of more advanced hepatic disease. Serum transaminases were monitored at baseline and once weekly for the duration of the study to permit a better understanding of the time course of potential improvement in hepatic inflammation during the course of this short study.
Time Frame: Baseline and Week 4
Population: The AST Population consists of all participants who received at least one dose of the study drug. One participant in the Placebo group did not have AST data for Day 28.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | MK-4074 | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 10 | 9
Percent change | -6.74 [-19.73 to 6.24] | -13.95 [-26.93 to -0.97] | -3.28 [-16.64 to 10.08]
Statistical Analysis 1: Comparison: MK-4074 vs Placebo; Test type: Superiority or Other; p > 0.200, Linear mixed effects model; Containing fixed effects for treatment, and predose Day 1 (baseline) as a fixed covariate; Least squares mean difference = -3.47, 95% CI 2-sided [-17.85 to 10.92]
Statistical Analysis 2: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p > 0.200, Linear mixed effects model; Containing fixed effects for treatment, and predose Day 1 (baseline) as a fixed covariate; Least squares mean difference = -10.67, 95% CI 2-sided [-25.06 to 3.71]

4. Primary Outcome: Number of Participants Experiencing One or More Adverse Events (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 10 weeks
Population: All Subjects as Treated (AST) Population consists of all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | MK-4074 | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Participants | 4 | 4 | 5

5. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 4
Time Frame: Up to 4 weeks
Population: The AST Population consists of all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | MK-4074 | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: The AST Population (Safety Population) consists of all participants who received at least one dose of the study drug.
Groups:
- Placebo for MK-4074: Participants will receive oral doses of placebo matching MK-4074 twice daily for 4 weeks.
- Pioglitazone: Participants will receive oral doses of pioglitazone hydrochloride 30 mg once daily for 4 weeks.
Arm/Group | MK-4074 | Placebo for MK-4074 | Pioglitazone | Placebo for Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 4/10 | 1/5 | 4/10 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4074 (N=10) | Placebo for MK-4074 (N=5) | Pioglitazone (N=10) | Placebo for Pioglitazone (N=5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.